CLINICAL TRIAL: NCT05258552
Title: Efficacy and Safety of Preoperative Enema in the Prevention of Catheter Dysfunction in Peritoneal Dialysis: A RCT Study
Brief Title: Efficacy of Preoperative Enema in the Prevention of Catheter Dysfunction in Peritoneal Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shiren sun, director of nephrology, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: enema for PD
Record Dates: First submitted 2022-02-09; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Peritoneal Dialysis Access Failure
MeSH Terms: interventions — Enema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enema group (Experimental)
  Interventions: Procedure: enema
- Control group (No Intervention)

INTERVENTIONS:
Procedure: enema — preoperative enema
  Arms: Enema group

SUMMARY:
A prospective, randomized, controlled study was conducted to identify patients with end-stage renal disease who required open peritoneal dialysis catheterization, preoperative enema or no enema was used to evaluate the efficacy and safety of reducing catheter dysfunction.

DETAILED DESCRIPTION:
A prospective, randomized, controlled study was conducted to identify patients with end-stage renal disease who required open peritoneal dialysis catheterization, preoperative enema or no enema was used to evaluate the efficacy and safety of reducing catheter dysfunction. All the patients were divided into two groups: preoperative enema group and no intervention group. The peritoneal dialysis malfuction were observed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18;
* Maintenance peritoneal dialysis treatment is required for end-stage Renal Disease;
* First-time open surgeon peritoneal dialysis catheterization patient;
* Only straight double-cuff Tenckhoff dialysis catheters were used.
* Willing to participate in this study and sign informed consent form.

Exclusion Criteria:

* peritoneal dialysis contraindication;
* Enema contraindication;
* Patients refuse enema;
* Expected survival time < 3 months;
* Catharsis such as Senna Leaf and lactulose used before operation or colonic dialysis and enema used 3 days before operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Catheter dysfunction requiring intervention within 3 months of peritoneal dialysis catheterization | 3 months
Time of first peritoneal dialysis catheter dysfunction | 6 months

SECONDARY OUTCOMES:
Incidence of Catheter dysfunction requiring intervention within 6 months of peritoneal dialysis catheterization | 6 months
Catheter survival time | 6 months
Incidence of peritoneal dialysis-associated Peritonitis | 6 months

IPD SHARING:
Plan to Share IPD: No